CLINICAL TRIAL: NCT04690244
Title: The Effect of Tai Chi Chuan on Cognitive and Motor Functions in Older Adults
Brief Title: The Effect of Tai Chi Chuan in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LithuanianSportsU-4
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Healthy Aging; Motor Learning; Cognitive Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi Chuan group (Experimental): Fifteen healthy elderly subjects participated in 10 weeks of Tai Chi Chuan practice. Inclusion criteria were:
  * aged 60 years and older;
  * sedentary behavior for at least 6 months;
  * no previous experience of Tai Chi Chuan practice;
  * good physical health determined by Physical Activity Readiness Questionnaire as - confirmed by medical history;
  * no cognitive impairments determined by baseline Mini-Mental State Examination score of ≥ 45.
  All participants were asked to not perform any sports activities while the research was ongoing.
  Interventions: Other: Tai Chi Chuan trainings
- Control group (No Intervention): In the control group, fifteen subjects also had to meet the same criteria and did not perform any exercises or make changes in their daily living life.

INTERVENTIONS:
Other: Tai Chi Chuan trainings — 10 weeks of Tai Chi Chuan practice by 6-year experienced training teacher, 2 times per week, 60 min per session.
  Arms: Tai Chi Chuan group

SUMMARY:
30 healthy older participants were enrolled in the study and were randomly classified into two groups. In the experimental group (n = 15) participants received 10-week Tai Chi Chuan practice intervention, in the control group (n=15) participants were asked do not change their living habits in 10 weeks. All participants had no practice Tai Chi Chuan before.

DETAILED DESCRIPTION:
All participants had to proceed with familiarization with cognitive function tests before all measurements and evaluation. Study protocol began in the early morning after overnight fasting (10.7 ± 4.7 h). Firstly, participants were asked to lay in the supine position for 15 minutes in rest to measure resting heart rate (HR) and heart rate variability (HRV) during the last 10 minutes and blood pressure afterward. Subsequently, participants completed PSS-10 and HADS questionnaires, and then a venous blood sample was taken for BDNF and irisin concentrations measurements. Then measurements of cognitive functions and motor learning were performed. After baseline assessments, participants were randomized to the experimental and control groups. The experimental group subjects (n=15; 13 women) participated in 10 weeks Tai Chi practice. In the control group, participants (n=15; 13 women) were instructed do not to engage in any additional sports practice. All tests and measurements were repeated after 10 weeks in the same order as it was at the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* age from 60 years old;
* voluntary participation in the study;
* does not have chronic diseases or injuries that may affect physical activity,
* does not have physical and mental disorders;
* has no hearing impairment;
* does not smoke;
* does not use psychotropic substances;
* pulse from 40 to 100 beats per minute at rest;
* impaired or corrected vision;
* blood pressure up to 139/89 mmHg at rest;
* never had practice of Tai Chi Chuan

Exclusion Criteria:

* persons suffering from: mental, oncological, cardiovascular, skeletal, muscular, respiratory disorders or diseases after physical exhaustion will not be invited to the study;
* after surgery; injuries (in last 3 years);
* contraindications to physical activity.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 10 weeks
  R-R intervals were recorded using a Polar H7 sensor with a chest strap (Kempele, Finland) in laying position, in rest.
Blood Pressure | 10 weeks
  Resting blood pressure was measured using digital electronic blood pressure monitor (Microlife BP A100, Widnau, Switzerland)
Perceived Stress Scale - PSS-10 | 10 weeks
  The purpose of this scale is to assess the degree of stress in subjects' lives. It consists of questions about the frequency of feeling and thoughts during the past time period. Potential answers: 0-never; 1-almost never; 2-sometimes; 3-fairly often and 4-very often. The scores are obtained by reversing the scores on the four positive items:for example, 0=4, 1=3, 2=2, etc. and then summing across all items. Scores for the 10-item form range from 0 to 40,with higher scores indicating greater perceived stress
Hospital Anxiety and Depression Scale (HADS) | 10 weeks
  To determine the level of anxiety and depression of subjects was used HADS scale. The scale consists of totally 14questions with the answers valued from 0 to 3. Half of questions addressed to estimate anxiety and rest - depression.The total scoring and conclusion for the both categories of questions: 0-7 = Normal; 8-10 = Borderline abnormal(borderline case); 11-21 = Abnormal (case)
Muscle circulatory BDNF Measurement | 10 weeks
  Venous blood samples from the median antecubital vein were collected in 5 ml vacuum tubes with a gel separator and was separated by centrifugation (15 min at 1200g) to make blood serum. Samples were aliquoted and stored at -20°C until analysis. The serum concentration of Human Free BDNF was measured using an enzyme-linked immunoassay kit(R&D Systems, Minneapolis, USA).
Circulating Irisin Measurement | 10 weeks
  Venous blood samples from the median antecubital vein were collected in 5 ml vacuum tubes with a gel separator and was separated by centrifugation (15 min at 1200g) to make blood serum. Samples were aliquoted and stored at -80°C until analysis. The serum concentration of Irisin was measured using a competitive ELISA, immobilized antigen immunoassay kit (BioVendor R&D Systems, Brno, Czech Republic).
Motor Learning Evaluation | 10 weeks
  The reaction time and velocity study will be measured with a DPA-1 analyzer. The DPA-1 device allows to study the reaction time, dynamic and kinematic characteristics of the movements.
Cognitive Function Performance Evaluation | 10 weeks
  The Automated Neuropsychological Assessment Metrics computer program, which assesses a person's neuropsychological condition, will be used to assess cognitive function indicators. Evaluates areas of cognition that are related to brain executive function. The following tests will be used in the study: Simple reaction time, Two choice reaction time, Memory search, Mathematical processing, Code substitution - learning, Code substitution - delayed, Go / No-Go, Matching grids.
Balance Evaluation | 10 weeks
  Balance measurement will be measured on a Kistler platform. The subjects' balance study evaluated static posturography using a force plate and computer equipment to record signals (KISTLER, Switzerland, Slimline System 9286). During the study, the subject stands on the force plate in four different positions.

SECONDARY OUTCOMES:
Weight Measurment | 10 weeks
  Body weight was measured by Tanita Body Composition Analyzer TBF-300 (Japan).
Height Measurement | 10 weeks
  The height was measured by a centimeter strip.

CONTACTS AND LOCATIONS:
Overall Officials: Rima Solianik, PhD, Principal Investigator — Lithuanian Sport University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No